CLINICAL TRIAL: NCT06822712
Title: A Prospective, Multicenter, Noninferiority, Randomized Controlled Clinical Trial Evaluating the Safety and Efficacy of Sirolimus-coated Coronary Balloon Dilatation Catheter vs Paclitaxel-coated Balloon Catheter for the Treatment of De Novo Coronary Bifurcation Lesions
Brief Title: Efficacy and Safety of Sirolimus-coated Coronary Balloon Dilatation Catheter for De Novo Coronary Bifurcation Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Collaborators: First Affiliated Hospital of Lanzhou University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM-D19-2
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-02

CONDITIONS: Coronary Arterial Disease (CAD)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Sirolimus-coated Coronary Balloon Dilatation Catheter
  Interventions: Device: Sirolimus-coated Balloon Dilatation Catheter
- Control Group (Active Comparator): Paclitaxel-coated Balloon Catheter (Brand: Bingo®)
  Interventions: Device: Paclitaxel-coated Balloon Dilatation Catheter

INTERVENTIONS:
Device: Sirolimus-coated Balloon Dilatation Catheter — During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using the Sirolimus-coated Balloon Dilatation Catheter in the test group, subsequently completing the remaining procedure
  Arms: Test Group
Device: Paclitaxel-coated Balloon Dilatation Catheter — During PCI, percutaneous transluminal coronary angioplasty is performed on the target lesion using the Paclitaxel-coated Balloon Dilatation Catheter in the control group, subsequently completing the remaining procedure
  Arms: Control Group

SUMMARY:
Evaluating the Safety and Efficacy of Sirolimus-coated Coronary Balloon Dilatation Catheter vs Paclitaxel-coated balloon catheter for the Treatment of De Novo Coronary Bifurcation Lesions

ELIGIBILITY:
Inclusion Criteria:

Participants in this clinical trial must meet all of the following criteria:

General Inclusion Criteria

1. Age ≥18 years and ≤80 years.
2. Evidence of asymptomatic myocardial ischemia, or stable/unstable angina, or myocardial infarction that occurred more than 7 days before enrollment and is now stable.
3. Suitable for any type of coronary artery revascularization, such as balloon angioplasty, stent implantation, and coronary artery bypass grafting (CABG).
4. Capable of understanding the purpose of the trial, willing to participate, and acknowledging the risks and benefits described in the informed consent document by signing the informed consent form, and willing to undergo invasive imaging follow-up.

Angiographic Inclusion Criteria

1. A maximum of 2 vessels requiring treatment, with no more than 3 lesions in total.
2. If the non-target lesion and the target lesion are in the same vessel, the non-target lesion must be located distal to the target lesion.
3. Successful interventional treatment of the non-target lesion prior to the target lesion.
4. Only one true bifurcation lesion requiring treatment (Medina classification 1.1.1, 1.0.1, 0.1.1), with a diameter stenosis ≥70% (by visual estimation) at the ostium of the target lesion side branch.
5. Successful pre-dilation/kissing balloon of the target lesion side branch, no dissection grade C or higher, residual stenosis ≤30% (by visual estimation) in the side branch lesion, and TIMI 3 flow.
6. Suitable for PCI, with the main branch lesion of the target lesion planned for stent implantation without drug-coated balloon treatment, and the side branch lesion treated with a drug-coated balloon without stent implantation; it is recommended to perform kissing balloon dilation for both the main and side branches.
7. Reference diameter of the target lesion side branch 2.0-4.0 mm, and lesion length ≤38 mm.

Exclusion Criteria:

If a participant has any of the following conditions, they will be excluded from the study:

General Exclusion Criteria

1. Unstable Arrhythmias: Such as high-risk ventricular premature beats or ventricular tachycardia.
2. Severe Heart Failure (New York Heart Association Functional Classification, NYHA Class IV).
3. Preoperative Renal Impairment: Or currently undergoing hemodialysis treatment.
4. Bleeding Tendencies or Contraindications to Antiplatelet Agents and Anticoagulants: Participants who cannot undergo antithrombotic therapy.
5. History of Peptic Ulcer or Gastrointestinal Bleeding within the Past 6 Months: Or history of cerebral hemorrhage, cerebral infarction, or other cerebrovascular accidents (stroke) within the past 6 months.
6. Known Allergies to Contrast Agents, Paclitaxel, Sirolimus, or Their Derivatives.
7. Life Expectancy Less Than 12 Months.
8. Poor Compliance: Participants who, in the investigator's judgment, are unlikely to adhere to the study requirements or are otherwise deemed unsuitable for inclusion.
9. Participation in Other Ongoing Clinical Trials: Participants who have not reached the primary endpoint in other ongoing clinical trials.
10. Pregnant or Lactating Women: Women who plan to conceive within 12 months or are unwilling to use effective contraception.

Angiographic Exclusion Criteria

1. Left Main Trunk and Its Bifurcation Lesions Requiring Treatment.
2. Thrombus in the Target Lesion: Excessive tortuosity of the vessel, making it unlikely for the balloon to pass through the lesion.
3. Total Occlusion in the Side Branch Lesion of the Target Lesion.
4. Severe Calcification in the Side Branch Lesion of the Target Lesion: Lesions that cannot be pre-dilated or treated with double-balloon kissing dilation.
5. In-Stent Restenosis in the Target Vessel (Including Both Main and Side Branches).
6. Residual Stenosis >30% (by Visual Estimation) or Dissection Grade C or Higher After Pre-Dilation or Double-Balloon Kissing Dilation of the Side Branch Lesion of the Target Lesion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Degree of stenosis | 9 Months postoperatively
  Degree of stenosis (%) of target bifurcation lesion segment diameter at 9 months postoperatively (Measured by QCA)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China